CLINICAL TRIAL: NCT06025773
Title: A Randomized, Open-label, 2x2 Crossover-design Clinical Trial to Evaluate the Safety and Pharmacokinetic/Pharmacodynamic Characteristics After Oral Administration of AD-212-A or AD-2121 in Healthy Adult Volunteers
Brief Title: A Study to Compare PK/PD Characteristics and Safety Profiles Between AD-212-A and AD-2121
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-212PK/PD-03
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole; Calcium Carbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): Period 1 : Reference Drug (AD-2121), Period 2 : Test Drug (AD-212-A)
  Interventions: Drug: Lansoprazole 15 mg; Drug: Lansoprazole 15mg/Calcium carbonate 600mg
- Arm-B (Experimental): Period 1 : Test Drug (AD-212-A), Period 2 : Reference Drug (AD-2121)
  Interventions: Drug: Lansoprazole 15 mg; Drug: Lansoprazole 15mg/Calcium carbonate 600mg

INTERVENTIONS:
Drug: Lansoprazole 15 mg — AD-2121 (Lansoprazole 15 mg), Oral, Capsule
Drug: Lansoprazole 15mg/Calcium carbonate 600mg — AD-212-A (Lansoprazole 15mg/Calcium carbonate 600mg), Oral, Tablet

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic and pharmacodynamic characteristics of AD-212-A in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic and pharmacodynamic characteristics and safety profiles of AD-212-A compared with AD-2121 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg and Body mass index (BMI) between 18.5 kg/m2 and 27.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit
* Negative result from Serum Helicobacter pylori antibody at the time of screening visit

Exclusion Criteria:

* Patients with trouble performing Gastric pH monitoring

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve over a dosing interval at steady state (AUCτ,ss) | pre-dose to 24 hours of 1st administration versus pre-dose to 24 hours of repeated administration (7days)
  AUCτ,ss after 7days repeated administration of Lansoprazole
Percent Decrease from baseline of Integrated gastric acidity | 24 hours before 1st administration to 24 hours after repeated administration (7days)
  Percent Decrease from baseline of Integrated gastric acidity after repeated adadministration of Lansoprazole
  Integrated gastric acidity calculation:
  (Integrated gastric acidity Before - Integrated gastric acidity after)/Integrated gastric acidity Before*100
  * Acid concentration (mM) = 1000 ⅹ 10-pH
  * Acidity (mmol.h/L) = (acid in mM at time 't' + acid in mM at time 't-1')/2 ⅹ (t-(t-1))
  * Integrated Acidity means cumulative sum per second for 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea